CLINICAL TRIAL: NCT03032419
Title: Safety and Immunogenicity of Adjuvanted Reduced Dose Inactivated Polio Vaccine, IPV-Al SSI, in Comparison to Non-adjuvanted Full Dose IPV SSI, in Infants Vaccinated at 6, 10, 14 Weeks and 9 Months of Age
Brief Title: Safety and Immunogenicity of Adjuvanted Reduced Dose Inactivated Polio Vaccine Given at 6, 10, 14 Weeks and 9 Months
Acronym: VIPV-06
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Larix A/S (Industry); Syneos Health (Other); AJ Vaccines A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VIPV-06
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPV-Al SSI (Experimental): IPV-Al contains the reduced dose of IPV to be administered intramuscularly to the anterolateral aspect of the right thigh. Each subject randomised to this group will receive three primary injection at 6, 10, and 14 weeks of age and one booster injection at 9 months of age
  Interventions: Biological: IPV-Al SSI
- IPV SSI (Active Comparator): IPV SSI contains the full dose of IPV to be administered intramuscularly to the anterolateral aspect of the right thigh. Each subject randomised to this group will receive three primary injection at 6, 10, and 14 weeks of age and one booster injection at 9 months of age
  Interventions: Biological: IPV SSI

INTERVENTIONS:
Biological: IPV-Al SSI — 3 primary injections of IPV-Al SSI at 6, 10, and 14 weeks of age and 1 booster at 9 months of age
  Arms: IPV-Al SSI
Biological: IPV SSI — 3 primary injections of IPV SSI at 6, 10, and 14 weeks of age and 1 booster at 9 months of age
  Other Names: IPV Vaccine SSI
  Arms: IPV SSI

SUMMARY:
The trial is a phase III, non-inferiority, observer-blind, randomised, controlled, multicentre clinical trial with 2 parallel groups: IPV-Al SSI (investigational vaccine) and IPV SSI (reference vaccine)

DETAILED DESCRIPTION:
In addition to the trial vaccine (IPV-Al SSI or IPV SSI), the trial subjects will receive vaccinations with the Philippine national childhood vaccination programme. The trial vaccine (IPV-Al SSI or IPV SSI) is administered in the RIGHT thigh, where other injectable childhood vaccines are administered in the opposite (LEFT) thigh. There are 6 trial visits:

Visit 1 (screening, 1st vaccination and blood sampling visit): written informed consent is obtained. Information on medical history, demographics and concomitant medication is collected, a physical examination is performed and the subject's eligibility is assessed according to the pre-specified in-/exclusion criteria. A pre-vaccination blood sample is taken for polio antibody measurements, and the subject is randomly allocated into one of the 2 groups and vaccinated. If it is not possible to draw a blood sample on Visit 1 the child cannot continue in the trial. The subject is observed for immediate AEs ½ an hour after all vaccinations. A diary, a ruler and a thermometer are handed out to the parents to record daily the temperature and injection site reactions, during the first 3 days after the vaccinations until resolved and to record any AEs as instructed by the trial staff. 2 days after Visit 1 the trial staff will make a telephone call to the parent(s)/guardian(s) to clarify any questions regarding the AE recording in the diary.

Visit 2 (2nd vaccination visit), 28-42 days after Visit 1: contraindications are reviewed, the 2nd vaccination is given, the diary is collected and AEs and concomitant medications (CMs) are recorded. A new diary is handed out.

2 days after Visit 2 the trial staff will make a telephone call to the parent(s)/guardian(s) to clarify any questions regarding the AE recording in the diary.

Visit 3 (3rd vaccination visit), 28-42 days after Visit 2: contraindications are reviewed, the 3rd vaccination is given, the diary is collected and AEs and CMs are recorded. A new diary is handed out. 2 days after Visit 3 the trial staff will make a telephone call to the parent(s)/guardian(s) to clarify any questions regarding the AE recording in the diary.

Visit 4 (blood sample visit), 28-42 days after Visit 3: a blood sample for polio antibody measurements is taken, the diary is collected, and AEs and CMs are recorded.

Visit 5 (4th vaccination and blood sample visit), at 9 months of age (+14 days): a blood sample is taken for polio antibody measurements, contraindications are reviewed, the 4th vaccination is given, and AEs and CMs are recorded. A new diary is handed out. 2 days after Visit 5 the trial staff will make a telephone call to the parent(s)/guardian(s) to clarify any questions regarding the AE recording in the diary.

Visit 6 (blood sample and end of trial visit), 28-42 days after Visit 5: a blood sample for polio antibody measurements is taken, the diary is collected, and AEs and CMs are recorded. The end of trial form is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Infants of 6 weeks of age (-3 to +14 days) on the date of the 1st vaccination
2. Healthy assessed from medical history and physical examination
3. Parent(s)/guardian(s) willing to let their infant follow the national Philippine childhood vaccination programme and schedule, in addition to let their infant receive the trial vaccine
4. Parent(s)/guardian(s) properly informed about the trial and has signed the informed consent form
5. Parent(s)/guardian(s) granting access to the infant's trial related medical records
6. Parent(s)/guardian(s) likely to comply with the trial procedures

Exclusion Criteria:

1. Vaccinated with any polio vaccine other than the trial vaccines, prior to inclusion or planned during the trial
2. OPV vaccination or known exposure to poliovirus (wild or vaccine derived) in household (living together) within 3 months prior to inclusion or planned during the trial
3. Low birth weight (< 2,500 g)
4. Known or suspected immunodeficiency (e.g. leukaemia, lymphoma) or family history of congenital or hereditary immunodeficiency. HIV infection is not an exclusion criteria
5. Severe uncontrolled chronic (e.g. neurologic, pulmonary, gastrointestinal, hepatic, renal or endocrine) disease
6. Known or suspected allergy to vaccine constituents (e.g. hypersensitivity to formaldehyde, aluminium or 2-phenoxyethanol)
7. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections or blood sampling
8. Treatment with a product which is likely to modify the immune response (e.g. blood products and immunoglobulins) prior to inclusion or planned during the trial
9. Participating in another clinical trial
10. Not suitable for inclusion in the opinion of the investigator

Ages: 6 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1002 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion for poliovirus type 1, 2 and 3 for IPV-Al compared to IPV SSI | Change from baseline to one month after 3rd vaccination

SECONDARY OUTCOMES:
Adverse event following vaccinations (key secondary) | After primary injections at 2, 4 and 6 months of age
Subjects with seroprotection against poliovirus types 1, 2 and 3 | One months after 3rd vaccination
Subjects with seroprotection against poliovirus types 1, 2 and 3 | Before and one month after the 4th vaccination
Subjects with poliovirus types 1, 2 and 3 post-vaccination titres ≥ 4-fold above the estimated titre of maternal antibody | One months after 3rd vaccination
Geometric mean titres (GMTs) and medians for poliovirus types 1, 2 and 3 | One months after 3rd vaccination
Geometric mean titres (GMTs) and medians for poliovirus types 1, 2 and 3 | Before and one month after the 4th vaccination
Reverse cumulative titre distribution curves for poliovirus types 1, 2 and 3 | From baseline, one month after 3rd vaccination, and before and one month after 4th vaccination

OTHER OUTCOMES:
Sensitivity analysis: subjects with ≥ 4-fold increases in poliovirus types 1, 2 and 3 titres | From baseline to one month after 3rd vaccination
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - seroprotection against poliovirus types 1, 2 and 3 | One month after 3rd vaccinations
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - seroprotection against poliovirus types 1, 2 and 3 | Before and one month after 4th vaccination
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - post-vaccination titre ≥ 4-fold above maternal titre against poliovirus types 1, 2 and 3 | One month after 3th vaccination
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - geometric mean titres and median for poliovirus types 1, 2 and 3 | One month after 3th vaccination
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - geometric mean titres and median for poliovirus types 1, 2 and 3 | Before and one month after 4th vaccination
Sensitivity analysis: sub-groups of infants with and without seroprotection at baseline - reverse cumulative titre distribution curves for poliovirus types 1, 2 and 3 | From baseline to one month after 4th vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kromann, Study Director — Statens Serum Institut
Locations (1):
- 5 sites in Philippines, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bravo LC, Carlos JC, Gatchalian SR, Montellano MEB, Tabora CFCB, Thierry-Carstensen B, Tingskov PN, Sorensen C, Wachmann H, Bandyopadhyay AS, Nielsen PI, Kusk MV. Immunogenicity and safety of an adjuvanted inactivated polio vaccine, IPV-Al, compared to standard IPV: A phase 3 observer-blinded, randomised, controlled trial in infants vaccinated at 6, 10, 14 weeks and 9 months of age. Vaccine. 2020 Jan 16;38(3):530-538. doi: 10.1016/j.vaccine.2019.10.064. Epub 2019 Nov 5. PMID 31703934